CLINICAL TRIAL: NCT06347991
Title: Alberta Chiropractic SelfBack Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Chiropractic Association of Alberta (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00140155
Record Dates: First submitted 2024-03-17; First posted 2024-04-04 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Those who receive the SelfBack app
  Interventions: Behavioral: SelfBack

INTERVENTIONS:
Behavioral: SelfBack — The SelfBack app is a promising decision support system (DSS) App used globally to support and reinforce desired self-management behavior for LBP. Selfback's program goal is to improve the self-management of nonspecific LBP to reduce pain-related disability.

SUMMARY:
Recurrent and persistent low back pain (LBP) is a massive problem in Canada that causes a substantial pain, disability, cost, and even premature death.

The good news is that treatments for recurrent and persistent LBP are available. Many guidelines now recommend education and exercise as the best intervention for chronic LBP. Unfortunately, education and exercise programs are not publicly funded in Canada-only Canadians with extended health benefits can access these programs.

As a result, the 50% of Canadians who do not have extended health benefits often seek care for LBP from their publicly funded physicians. Physicians, in turn, have little choice but to reach for what they have available, including opioids, x-rays and referrals to specialists. Not only are these interventions unhelpful for chronic LBP, they are often harmful, sometimes deadly, and disproportionately affect lower socio-economic status households.

A possible solution to this problem exists in a validated app (SelfBack) that provides tailored self-management plans consisting of advice on physical activity, physical exercises, and educational content. Tailoring of treatment plans to individuals is achieved by using case-based reasoning (CBR) methodology which is a branch of artificial intelligence.

This study will evaluate the feasibility of distributing the SelfBack app to persons experiencing LBP through their chiropractors.

The results of this study will help us understand the barriers and facilitators of distributing and using the app through Alberta Chiropractors. This information will be used to apply for funding for a larger study to understand the effectiveness of the app as an intervention for persistent and recurrent LBP.

DETAILED DESCRIPTION:
Purpose

This study will evaluate the feasibility of distributing the SelfBack app through members of the Chiropractic Association of Alberta and the feasibility of patients using the app.

Justification

The SelfBack app is a promising decision support system (DSS) App used globally to support and reinforce desired self-management behaviour for LBP. Selfback's program goal is to improve the self-management of nonspecific low back pain (LBP) to reduce pain-related disability. Using applications (apps) has been suggested to be a promising way to increase the effectiveness of self-management interventions.

Objectives

Our primary objective is to evaluate the feasibility of distributing and using the SelfBack app. A secondary objective is to assess patient outcomes collected by the SelfBack app.

Methodology Overview

The Chiropractic Association of Alberta (CAA) will recruit members who are interested in being enrolled in the study. Those who meet the eligibility criteria and provide consent will then be trained in the SelfBack app and then respond to a baseline survey to determine their current attitudes and beliefs regarding using the SelfBack app. Trained and enrolled chiropractors will then identify chronic LBP patients in their own practice to receive the SelfBack App. Patients who are eligible and consent to participate will be provided with the SelfBack App. The SelfBack app then collects patient data and provides patients with personalized advice regarding education and exercise for chronic LBP. De-identified group-level Selfback data will then be downloaded by the investigative team at regular intervals for analysis. Finally, chiropractors will provided with a follow-up survey to evaluate their attitudes and beliefs following their involvement in the trial.

Overall timeline and setting:

The study will occur between May 2024 and December 2024 (8 months).

Patient Data

Once patients provide consent to the Investigative Team, they will be sent instructions on how to download and use the SelfBack app. Once installed on the participant's smartphone, the SelfBack app will ask a series of baseline questions (~ 30 min) to establish what educational advice and exercises best suit the participant.

The SelfBack app regularly asks questions of the user to determine their ability to participate in exercise and education and evaluate their progress in the program. The list of survey questions used by the app was created, approved, and distributed by Selfback and is attached to this protocol.

The SelfBack will collect two categories of data.

The first category will be related to patient demographics.

The second category is related to patient-related outcome measures, a variety of established scales, and questionnaires with known psychometric properties. These outcome measures are used to assess the participant's health status, fitness level, and psychological health. These specific outcomes are asked at baseline, 3, and 6 months.

Clinician - Patient Interaction

Chiropractors are not excluded from seeing their patients while patients are using the SelfBack app. Clinical encounters may occur for heart concerns that are unrelated to the study or require in-person evaluation to determine and evaluate their ability to continue in the study.

Clinicians are also provided with a real-time dashboard through Selfback where they can receive information about SelfBack users in real-time. Specifically, the dashboard shows if triggers have occurred which indicates the patient has entered information into the app which requires monitoring or follow-up.

Analyses

The general procedure for statistical analysis is as follows:

Descriptive statistics will be generated which will be cross-tabulated with demographic groups of interest (e.g., gender, age, community size, caregiver status, self-identification of disability, and ethnic and racial identification).

Feasibility will be judged as successful if 50% of the enrolled participants complete the education and exercise program recommended by the app.

ELIGIBILITY:
Clinician Inclusion Criteria:

* Practicing chiropractor in Alberta.
* Will have access to ATLAS, ChiroSUITE, or Jane software packages
* Must have completed and filed a Privacy Impact Assessment with the Government of Alberta, as identified under the Health Information Act.
* Connected to Alberta's electronic health record, Netcare

Patient Inclusion Criteria:

* Patients of enrolled chiropractors having persistent and/or recurrent LBP defined as those currently having LBP that has impacted daily activities for > 1 month. I
* Alberta resident 18 years of age or older
* Must have a personal smartphone with internet access.
* Must have a working e-mail address.
* Must speak, read, and write English or have regular access to persons who can assist in this regard.

Patient exclusion criteria:

* Patients who have complex back pain that requires direct clinical oversight.
* Patients with cognitive impairments or learning disabilities that limit participation.
* Patients with serious mental illness.
* Patients who have non-LBP illnesses or conditions that are contraindicated to participation in SelfBack (e.g. exercise).
* Patients who have terminal illness
* Patients who are unable to take part in exercise/physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who utilize the SelfBack app | 8 months
  Success will be defined as 50% of patients using the app

SECONDARY OUTCOMES:
The percentage of clinicians who utilize the SelfBack app | 8 months
  Success will be defined as 50% of clinicians using the app

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No